CLINICAL TRIAL: NCT00564447
Title: A Single-Center, Open-Label, Randomized Study of the Pharmacokinetics of AzaSite Ophthalmic Solution Versus Vigamox in the Conjunctiva of Healthy Volunteers Following a Single Ocular Administration
Brief Title: Study of AzaSite (Azithromycin) Versus Vigamox in the Conjunctiva of Healthy Volunteers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Saiid Davari, Inspire Pharmaceuticals, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 041-102; P08654
Record Dates: First submitted 2007-11-20; First posted 2007-11-28 (Estimated); Results first posted 2011-07-26 (Estimated); Last update posted 2011-09-22 (Estimated); Status verified 2011-09

CONDITIONS: Bacterial Infections; Eye Infections
MeSH Terms: conditions — Bacterial Infections; Eye Infections | interventions — Azithromycin; Moxifloxacin

ARMS (8):
- Azithromycin-30 minutes Post dose (Experimental)
  Interventions: Drug: Azithromycin
- Azithromycin-2 hours post dose (Experimental)
  Interventions: Drug: Azithromycin
- Azithromycin-12 hours post dose (Experimental)
  Interventions: Drug: Azithromycin
- Azithromycin-24 hours post dose (Experimental)
  Interventions: Drug: Azithromycin
- Moxifloxacin-30 minutes post dose (Experimental)
  Interventions: Drug: Moxifloxacin
- Moxifloxacin-2 hours post dose (Experimental)
  Interventions: Drug: Moxifloxacin
- Moxifloxacin-12 hours post dose (Experimental)
  Interventions: Drug: Moxifloxacin
- Moxafloxacin-24 hours post dose (Experimental)
  Interventions: Drug: Moxifloxacin

INTERVENTIONS:
Drug: Azithromycin — azithromycin topical solution 1% given as a single drop in a single eye
  Other Names: AzaSite
  Arms: Azithromycin-12 hours post dose; Azithromycin-2 hours post dose; Azithromycin-24 hours post dose; Azithromycin-30 minutes Post dose
Drug: Moxifloxacin — Moxifloxacin topical solution given as a single drop in a single eye
  Other Names: Vigamox
  Arms: Moxafloxacin-24 hours post dose; Moxifloxacin-12 hours post dose; Moxifloxacin-2 hours post dose; Moxifloxacin-30 minutes post dose

SUMMARY:
The purpose of this study is to evaluate the drug concentrations of AzaSite™ compared to Vigamox at various time points in conjunctiva tissue of healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

* Have best corrected visual acuity of 0.60 logMAR or better in each eye as measured using Early Treatment of Diabetic Retinopathy Study chart

Exclusion Criteria:

* Have a known allergy and/or sensitivity to the test article(s) or its components or any therapies associated with the trial
* Have active signs or symptoms of any clinically significant ocular disorder (other than refractive disorders)
* Have a known bleeding disorder or history of bleeding complications after surgical or dental procedures
* Take aspirin, or take any other blood thinners or anti-coagulants (e.g. warfarin) including prescription, over the counter, or homeopathic therapies
* Have undergone any ocular surgical intervention within 3 months prior to Visit 1 or anticipate having ocular surgery during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2007-12; Primary Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Reza Haque, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Derived] Torkildsen G, O'Brien TP. Conjunctival tissue pharmacokinetic properties of topical azithromycin 1% and moxifloxacin 0.5% ophthalmic solutions: a single-dose, randomized, open-label, active-controlled trial in healthy adult volunteers. Clin Ther. 2008 Nov;30(11):2005-14. doi: 10.1016/j.clinthera.2008.10.020. PMID 19108788

RESULTS

PARTICIPANT FLOW:
Recruitment Details: December 2007
Pre-assignment Details: Normal volunteers
Period: Overall Study
Arm/Group | Azithromycin Ophthalmic Solution, 1% -30 Minutes Post Dose | Azithromycin Ophthalmic Solution, 1% -2 Hours Post Dose | Azithromycin Ophthalmic Solution, 1% -12 Hours Post Dose | Azithromycin Ophthalmic Solution, 1% -24 Hours Post Dose | Moxifloxacin 0.5% Ophthalmic Solution-30 Minutes Post Dose | Moxifloxacin 0.5% Ophthalmic Solution-2 Hours Post Dose | Moxifloxacin 0.5% Ophthalmic Solution-12 Hours Post Dose | Moxifloxacin 0.5% Ophthalmic Solution-24 Hours Post Dose
Started | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Azithromycin Ophthalmic Solution, 1% -30 Minutes Post Dose | Azithromycin Ophthalmic Solution, 1% -2 Hours Post Dose | Azithromycin Ophthalmic Solution, 1% -12 Hours Post Dose | Azithromycin Ophthalmic Solution, 1% -24 Hours Post Dose | Moxifloxacin 0.5% Ophthalmic Solution-30 Minutes Post Dose | Moxifloxacin 0.5% Ophthalmic Solution-2 Hours Post Dose | Moxifloxacin 0.5% Ophthalmic Solution-12 Hours Post Dose | Moxifloxacin 0.5% Ophthalmic Solution-24 Hours Post Dose | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 48
Age Continuous [Mean (Standard Deviation); unit: years] | 44.5 (11.1) | 46.8 (13.1) | 38.2 (13.2) | 33.7 (16.8) | 43.0 (13.7) | 43.5 (13.2) | 33.3 (8.2) | 36.7 (11.7) | 40.0 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 2 | 3 | 1 | 5 | 2 | 3 | 23
  Male | 1 | 4 | 4 | 3 | 5 | 1 | 4 | 3 | 25
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 48

OUTCOME MEASURES:

1. Primary Outcome: Assessment of Pharmacokinetic Parameters
Time Frame: Up to 24 hours
Reporting Status: Not Posted

2. Primary Outcome: Assessment of Pharmacokinetic Parameters
Description: Conjunctiva Concentration of Azithromycin and Moxifloxacin
Time Frame: Over 24 hours
Measure: Mean (Standard Deviation); unit: μg/g
Arm/Group | Azithromycin Ophthalmic Solution, 1% -30 Minutes Post Dose | Azithromycin Ophthalmic Solution, 1% -2 Hours Post Dose | Azithromycin Ophthalmic Solution, 1% -12 Hours Post Dose | Azithromycin Ophthalmic Solution, 1% -24 Hours Post Dose | Moxifloxacin 0.5% Ophthalmic Solution-30 Minutes Post Dose | Moxifloxacin 0.5% Ophthalmic Solution-2 Hours Post Dose | Moxifloxacin 0.5% Ophthalmic Solution-12 Hours Post Dose | Moxifloxacin 0.5% Ophthalmic Solution-24 Hours Post Dose
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
μg/g | 130.8 (89.1) | 51.6 (26.0) | 67.1 (51.8) | 31.9 (20.4) | 1.9 (2.0) | 3.8 (9.0) | 0.0 (0.0) | 0.0 (0.0)

ADVERSE EVENTS:
Arm/Group | Azithromycin Ophthalmic Solution, 1% -30 Minutes Post Dose | Azithromycin Ophthalmic Solution, 1% -2 Hours Post Dose | Azithromycin Ophthalmic Solution, 1% -12 Hours Post Dose | Azithromycin Ophthalmic Solution, 1% -24 Hours Post Dose | Moxifloxacin 0.5% Ophthalmic Solution-30 Minutes Post Dose | Moxifloxacin 0.5% Ophthalmic Solution-2 Hours Post Dose | Moxifloxacin 0.5% Ophthalmic Solution-12 Hours Post Dose | Moxifloxacin 0.5% Ophthalmic Solution-24 Hours Post Dose
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 1/6 | 1/6 | 1/6 | 0/6 | 3/6 | 2/6 | 0/6 | 1/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Azithromycin Ophthalmic Solution, 1% -30 Minutes Post Dose (N=6) | Azithromycin Ophthalmic Solution, 1% -2 Hours Post Dose (N=6) | Azithromycin Ophthalmic Solution, 1% -12 Hours Post Dose (N=6) | Azithromycin Ophthalmic Solution, 1% -24 Hours Post Dose (N=6) | Moxifloxacin 0.5% Ophthalmic Solution-30 Minutes Post Dose (N=6) | Moxifloxacin 0.5% Ophthalmic Solution-2 Hours Post Dose (N=6) | Moxifloxacin 0.5% Ophthalmic Solution-12 Hours Post Dose (N=6) | Moxifloxacin 0.5% Ophthalmic Solution-24 Hours Post Dose (N=6)
Conjunctival Haemorrhage (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Eyelid Margin Crusting (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Eye Pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other